CLINICAL TRIAL: NCT05914207
Title: Effects of Lifestyle Modifications and Vestibular Rehabilitation Therapy in Children and Adolescents With Vestibular Migraine
Brief Title: Non-Pharmacological Treatment of Vestibular Migraine in Children and Adolescent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Jeyasakthy Saniasiaya, Principal Investigator, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MECID.No 2023224-12175
Record Dates: First submitted 2023-05-08; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Vestibular Migraine
Keywords: Children; Adolescent; Non-pharmacological; lifestyle modifications; vestibular rehabilitation therapy

STUDY DESIGN:
Intervention Model Description: Children and adolescents who are diagnosed with Vestibular Migraine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vestibular Migraine group (Experimental): Written, verbal and pictorial descriptions will be provided for each participant regarding lifestyle modifications and vestibular rehabilitation exercise
  Interventions: Behavioral: Lifestyle modifications; Other: Vestibular rehabilitation exercise

INTERVENTIONS:
Behavioral: Lifestyle modifications — Written suggestions on lifestyle modifications including duration of sleep, meal frequency, reduce screen time, exercise duration, food to avoid.
Other: Vestibular rehabilitation exercise — Each participant will be taught simple home-based vestibular rehabilitation exercise, which needs to be repeated

SUMMARY:
Vestibular dysfunction has traditionally been linked to various conditions that affect older adults. Recent studies have shown that children and adolescents suffer from vestibular impairments, yet the numbers are still low due to some factors, including the non-typical presentations. Vestibular migraine has been found to be the most common condition of vestibular dysfunction among children and adolescents. Nonetheless, most children remain undiagnosed due to lack awareness and vague clinical presentations. Parallel to that, there has been no consensus regarding the management algorithm. Most children are managed with pharmacological management extrapolated from the adult algorithm. Many clinicians fail to understand that pharmacological treatments are not sustainable long-term and should focus on lifestyle modifications such as sleep and dietary habits and other non-pharmacological treatments such as deep breathing exercises and vestibular rehabilitation therapy. This study aims to investigate the effect of non-pharmacological treatment in managing children and adolescents with VM. The investigators will use a standardised questionnaire before and after interventions to investigate the effect of lifestyle modifications, simple vestibular rehabilitation exercises and deep breathing techniques in children and adolescents with VM. Lifestyle modifications and vestibular rehabilitation exercise is a more sustainable way of managing children and adolescents with VM, avoiding the side effects of medication, and is more cost-effective. If the non-pharmacological treatment shows promising results, the investigators will continue with multicentre randomised-controlled studies.

DETAILED DESCRIPTION:
The prevalence of vestibular dysfunction is approximately 30.4% among children and adolescents. Yet, the exact prevalence in children remains a quandary owing to several factors: difficulties describing symptoms and cannot differentiate between true vertigo, unsteadiness, imbalance and light-headedness; secondly, the short-lived nature of some peripheral vestibular conditions results in early and rapid compensation; thirdly, nuanced clinical manifestations of vestibular as well as balance impairment accounts for it being overlooked finally, lack of specialists to manage children with vestibular impairment.

Vestibular dysfunction or impairment results in disturbance in the body's balance system. Nonetheless, the most common symptoms include vertigo, nausea, vomiting, intolerance to head motion, nystagmus, unsteady gait, and postural instability. Although clinical presentation may be mild, vestibular dysfunction may impact the quality of life and day-to-day activity, especially school activities such as reading and learning, which are vital for these age groups.

Vestibular loss affects cognitive and emotional disturbance related to reflexive deficits, which are related to the role of ascending vestibular pathway to the limbic system and the neocortex's role in the sense of spatial orientation. Vestibular and balance impairment amongst adolescents and young adults will, in the long term, affect social, emotional, psychological and quality of life as vestibular and balance function is imperative in day-to-day life and activity.

Vestibular migraine (VM) is found to be the most common cause of dizziness among children and adolescents. The exact prevalence of VM remains unknown as VM is still underdiagnosed due to a lack of awareness amongst parents and attending physicians. It is worth noting that the diagnosis of VM in children and adolescents has traditionally been based on the description of clinical symptoms by the patient or parents/caretaker. The lack of definitive biomarkers and gold-standard diagnostic tools contributes to the delay in diagnosis. The typical battery of investigations, including otological, neurological, ophthalmological, and imaging performed, are oftentimes carried out to rule out other pathological disorders.

Vestibular migraine in children is diagnosed based on diagnostic criteria which recently has been put forth by the Committee for the Classification of Vestibular Disorders of the Bar any Society (ICVD) and the Migraine Classification subgroup of the International Headache Society, which describes the three spectrums of VM: Vestibular Migraine of Childhood, probable Vestibular Migraine of Childhood and Recurrent Vertigo of Childhood specific for children under 18 years of age.

No gold standard investigation tool exists to diagnose VM, as the available investigations are performed mainly to exclude other conditions such as Meniere's disease and BPPV.

Additionally, there is no evidence-based approach for treating VM in children and adolescents, with most recommendations extrapolated from reports on adult and childhood migraine headaches. Only two included studies described medication for VM. Overall, treatment for VM can be divided into pharmacological and non-pharmacological treatment. Pharmacological treatment of VM in children includes those taken during acute attacks and prophylactic treatment. Vestibular suppressants and triptans have been used to abort acute attacks in children and adolescents, although the exact efficacy is still unknown.

Non-pharmacological treatment aimed as a prophylactic measure such as eliminating migraine-triggering diet, vestibular rehabilitation, supplements, and a healthy lifestyle. Triggering factors such as increased screen time and usage of immersive technology needs attention parallel to getting adequate sleep, a healthy diet and breathing exercise. Lifestyle modifications have shown significant improvement among adult patients diagnosed with definite VM. Yet, no studies involving children and adolescents. The investigators aim to conduct a study to investigate the effect of lifestyle modifications, simple home-based vestibular rehabilitation and deep breathing exercise in children and adolescents diagnosed with VM. Lifestyle modifications, vestibular rehabilitation exercise and deep breathing exercise is a more sustainable way of managing children and adolescents with VM, avoids the side effects of medication, and is cost-effective.

Hypothesis The investigators hypothesise that non-pharmacological treatment which involves lifestyle modifications, home-based vestibular rehabilitation therapy and deep relaxation breathing, will be effective in controlling and reducing the symptoms of vestibular migraine in children and adolescents.

Innovation The majority of the studies on pharmacological interventions for vestibular migraine revolve around adult patients. Although the optimal treatment algorithm among adult vestibular migraine remains debatable, the effect of lifestyle modifications in vestibular migraine adult patients has shown promising results. The current research is innovative as the investigators will use an elaborate guide of lifestyle modifications which focuses on the child's dietary, sleep, and lifestyle habits, including increased physical activity, reduction of screen time as well as incorporating simple home-based vestibular rehabilitation therapy and deep breathing exercise. All children and adolescents will be diagnosed with vestibular migraine of childhood according to the Barany Consensus criteria. The investigators will divide the participants into 2 groups: children and adolescents. The investigators believe that the proposed investigation will be a more sustainable way to control, reduce vestibular migraine symptoms, and improve the overall quality of life among the participants. The findings from this research will be the foundation and pave the way for future larger-scale multicentre studies.

Research plan The investigators propose that an elaborate guide to lifestyle modifications focusing on the child's dietary, sleep, lifestyle habits, in addition to simple home-based vestibular rehabilitation therapy and deep breathing exercise, will reduce and improve vestibular symptoms in children and adolescents. No studies on non-pharmacological intervention among children and adolescents with vestibular migraine have been published. Yet, data involving adult patients have shown promising results, although no study involving adult patients with vestibular migraine has looked into the effect of lifestyle modifications which includes dietary and sleep habits, in addition to incorporating vestibular rehabilitation therapy and deep breathing exercise in a single study.

Justification of the study

Lifestyle modifications have successfully prevented Vestibular migraine (VM) in the adult study. No studies involving children and adolescents with VM have been carried out. The investigators aim to conduct a study to investigate the effect of lifestyle modifications and simple vestibular rehabilitation in children and adolescents diagnosed with VM. Lifestyle modifications and vestibular rehabilitation exercise is a more sustainable way of managing children and adolescents with VM, avoiding the side effects of medication and being cost-effective.

It is important to investigate the effects of lifestyle modifications on VM because the underlying causes of vestibular migraine are unclear. Our modifications include food triggers, restful sleep, exercise, eating regularity, vestibular rehabilitation, and deep breathing exercise. The investigators hypothesize comprehensive lifestyle modifications, vestibular rehabilitation, and deep breathing exercise will improve vestibular migraine symptoms. This project is important because vestibular migraine is reported to be one of the most common causes of vertigo, and interventions useful for other migraine types or vestibular symptoms may not be effective for VM in children and adolescents. If the investigators demonstrate improvement with comprehensive lifestyle modifications, the investigators will continue the line of investigation with randomized, controlled studies. This work furthers our goal of helping children and adolescents with VM.

Main Objective To investigate the effects of elaborate lifestyle modifications, vestibular rehabilitation therapy and deep breathing exercise among children and adolescents with vestibular migraine.

Specific Objective

* To determine the effect of lifestyle modifications, vestibular rehabilitation therapy and deep breathing exercise on the paediatric Dizziness Handicap Inventory (P-DHI)[5-12] and Dizziness Handicap Inventory (DHI) [13-18] pre and post-intervention
* To determine the effect of lifestyle modifications, vestibular rehabilitation therapy and deep breathing exercise on the overall quality of life pre and post-intervention

Hypothesis Comprehensive lifestyle modifications will improve the self-perceived impact of the symptoms of dizziness and headache in individuals with vestibular migraine.

Study endpoints

To determine the outcome of lifestyle modifications, vestibular rehabilitation and deep breathing exercises in children and adolescents with VM

Methodology

Study Type and Design

Study design: Exploratory Prospective cross-sectional study

* Duration: 2 years
* Subjects: Children and Adolescents aged between 5 to 18 years

Study population:

Patients aged between 5-18 years of age attending the Paediatric Vestibular and balance (ENT) clinic

Patients aged between 5 to 18 years old will be screened based on inclusion and exclusion criteria. Once the patient or parent/caretaker consents to participate in the study, the patient will be interviewed to complete a proforma, including the patient's socio-demographic, past medical history, otological, vestibular and balance complaints, and otoscopic examination. The patient, parent/caretaker will fill P-DHI or the DHI questionnaire at the first visit. This will be followed by a hearing assessment with pure tone audiometry and tympanometry, a routine examination for children and adolescents with vestibular symptoms. This will be followed by bedside vestibular assessment with video head impulse test (VHIT), cervical vestibular evoked myogenic potential (cVEMP), and subjective visual vertical (SVV). All test procedures were performed using a non-invasive technique and were explained to all participants before starting.

FLOWCHART

Patients aged 5-18 years fulfill the Barany criteria of VM

Socio-demographic, Otological, Vestibular Screening

1. st visit P-DHI (5-12yrs) or DHI (13-18)

   Lifestyle modifications + VRT regime
2. nd visit 4 weeks, 8 weeks: repeat P-DHI (5-12yrs) or DHI (13-18)

Study Population Children and adolescents aged between 5 to 18 years attending UMMC or in the community, either students in University Malaya or secondary school students in Klang Valley.

Withdrawal Criteria:

Subjects can choose to withdraw at any time. However, it is worth noting that all the investigations included in this study are safe.

Sample Size: 60 (Pilot study) Post-hoc power analysis will be done following data collection

Study Duration and Timeline: 2 years

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between 5-18 years
* Diagnosed with vestibular migraine based on the Diagnostic criteria consensus document of the Classification Committee of Vestibular Disorders of the Bárány Society and the International Headache Society

Exclusion Criteria:

* Not able to comprehend or able to follow instructions
* syndromic, other ontological, neurological conditions

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Paediatric Dizziness Handicap Inventory | This measure is carried after one month
  This measure assesses impact of dizziness in children between 5-12 years
Dizziness Handicap Inventory | This measure is carried out after one month
  This measure assesses impact of dizziness in children above 12 -18

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya Medical Centre, Kuala Lumpur, Malaysia